CLINICAL TRIAL: NCT06592794
Title: A Phase 3, Randomized, Observer-blinded, Placebo-controlled Study to Evaluate the Safety and Efficacy of mRNA-1403, a Multivalent Candidate Vaccine to Prevent Norovirus Acute Gastroenteritis in Adults ≥18 Years of Age
Brief Title: A Study to Investigate the Safety and Efficacy of mRNA-1403 in Participants ≥18 Years of Age for the Prevention of Acute Gastroenteritis
Acronym: Nova 301
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1403-P301
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Gastroenteritis; Norovirus Acute Gastroenteritis
Keywords: Acute Gastroenteritis; Norovirus Acute Gastroenteritis; mRNA-1403; Viral Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1403 (Experimental): Participants will receive a single injection of mRNA-1403 on Day 1.
  Interventions: Biological: mRNA-1403
- Placebo (Placebo Comparator): Participants will receive a single injection of mRNA-1403 matching placebo (0.9% sodium chloride solution) on Day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1403 — Intramuscular (IM) injection.
  Arms: mRNA-1403
Biological: Placebo — 0.9% sodium chloride solution by IM injection.
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to evaluate the safety and reactogenicity of mRNA-1403, and to demonstrate the efficacy of mRNA-1403 to prevent protocol-defined moderate or severe norovirus acute gastroenteritis (AGE) associated with vaccine matched genotypes.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who understand and are willing and physically able to comply with protocol mandated follow-up, including all procedures as assessed by the Investigator, and who are primarily responsible for their self-care and activities of daily living.
2. Participants may have chronic medical diagnoses but should be medically stable as assessed by the following criteria:

   * Absence of medical events associated with underlying diagnoses and qualifying as SAEs within 1 month prior to study intervention on Day 1.
   * Absence of known, current, and life-limiting diagnoses, which could continue for the duration of the study and which, in the opinion of the Investigator, would make completion of the protocol unlikely.
3. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
4. Participants assigned female at birth are eligible to participate if they are not pregnant or breastfeeding/chestfeeding/bodyfeeding and meet protocol defined criteria.

Exclusion Criteria:

1. Participant is acutely ill or febrile (temperature ≥38.0 degrees Celsius (°C) [100.4 degrees Fahrenheit [°F]) 72 hours prior to or at the Screening Visit or Day 1.
2. History of AGE within 14 days prior to Day 1 or close contact with an individual with AGE symptoms (in the home, socially, or occupationally) within 14 days prior to Day 1.
3. History of a diagnosis or condition that in the judgment of the Investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
4. Current diagnosis of chronic gastrointestinal (GI) disease that is associated with ongoing symptoms of regular vomiting and/or diarrhea. Participants with stable, well-controlled chronic GI disease without regular vomiting and/or diarrhea can be considered for enrollment.
5. Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation or that could interfere with safety assessments or interpretation of results according to the investigator's judgment.
6. Has undergone surgical procedures within 7 days prior to Day 1 or is scheduled to undergo a surgical procedure within 28 days after study intervention.
7. Reported history of congenital or acquired immunodeficiency, immunocompromising/immunosuppressive condition, asplenia, or recurrent severe infections per protocol.
8. Reported history of anaphylaxis, urticaria, or other significant AR requiring medical intervention after receipt of a vaccine or intervention that includes one or more of the same components contained in the study vaccine.
9. History of myocarditis, pericarditis, or myopericarditis with onset within 180 days prior to Day 1 whose values have not returned to Baseline clinical status.
10. History of Guillain-Barré syndrome.
11. Reported history of coagulopathy or bleeding disorder considered a contraindication to IM injection or phlebotomy.
12. Dermatologic conditions that could affect local solicited AR assessments.
13. Diagnosis of malignancy within the previous 2 years (excluding nonmelanoma skin cancer).
14. Has received systemic immunosuppressive therapies for >14 days in total within 6 months prior to Day 1 (for corticosteroids ≥10 milligrams (mg)/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
15. Has received or plans to receive any licensed vaccine ≤28 days prior to or within 28 days after study intervention (Day 1), except for influenza vaccines, which may be given 14 days before or after receipt of a study intervention.
16. Receipt of systemic immunoglobulins or blood products within 3 months prior to Day 1 or plans for receipt during the study.
17. Has donated ≥450 mL of blood products within 28 days prior to Day 1 Visit or plans to donate blood products during the study.
18. Participated in a clinical study with investigational treatment within 90 days prior to Day 1 (Baseline) based on the medical history interview or plans to do so while participating in this study. Participants may continue in prior interventional study follow-up activities, provided that it does not involve further investigational treatment and/or procedures that may affect safety and/or other study endpoints, and study participation does not result in a breach of either study protocol.
19. Is working as, has worked as, or is an immediate family member or household member of study personnel, Sponsor personnel, or study site staff directly involved with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28000 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Day 1 up to Day 7 (7 days after study intervention)
Number of Participants with Unsolicited Adverse Events (AEs) | Day 1 up to Day 28 (28 days after study intervention)
Number of Participants with Medically Attended Adverse Events (MAAEs) | Day 1 through Day 181
Number of Participants with Serious Adverse Events (SAEs), AEs of Special Interest (AESIs), and AEs Leading to Study Withdrawal | Day 1 up to Day 546 (Cohort 1) and Day 365 (Cohorts 2 and 3)
Vaccine Efficacy (VE) of mRNA-1403 to Prevent First Occurrence of Protocol-defined Moderate or Severe AGE Associated with Vaccine Matched Genotypes | Day 15 up to 6 months after the last participant dosed in each cohort

SECONDARY OUTCOMES:
VE of mRNA-1403 to Prevent First Occurrence of Protocol-defined Severe AGE Associated with Vaccine Matched Genotypes | Day 15 up to 6 months after the last participant dosed in each cohort
VE of mRNA-1403 to Prevent First Occurrence of Protocol-defined Severe Norovirus (NoV) AGE Associated with Any Genogroup I or II Norovirus (NoV) Genotype | Day 15 up to 6 months after the last participant dosed in each cohort
VE of mRNA-1403 to Prevent First Occurrence of Protocol-defined Moderate or Severe AGE Associated with Any Genogroup I or II NoV Genotype | Day 15 up to 6 months after the last participant dosed in each cohort
VE of mRNA-1403 to Prevent First Occurrence of Protocol-defined AGE of Any Severity Associated with Vaccine Matched NoV Genotypes | Day 15 up to 6 months after the last participant dosed in each cohort
VE of mRNA-1403 to Prevent Any Occurrence of Medically Attended AGE Associated with Vaccine Matched NoV Genotypes, as well as any Genogroup I or II NoV Genotype | Day 15 up to Day 546 (Cohort 1) and Day 365 (Cohorts 2 and 3)
VE of mRNA-1403 to Prevent Any Occurrence of AGE Hospitalizations Associated With Vaccine Matched NoV Genotypes, as well as any Genogroup I or II NoV Genotype | Day 15 up to Day 546 (Cohort 1) and Day 365 (Cohorts 2 and 3)
VE of mRNA-1403 to Prevent Any Occurrence of Protocol-defined Moderate or Severe AGE Associated with Vaccine Matched Genotypes | Day 15 up to Day 546 (Cohort 1) and Day 365 (Cohorts 2 and 3)
VE of mRNA-1403 to Prevent Any Occurrence of Protocol-defined AGE of Any Severity Associated with Any Genogroup I or II NoV Genotype | Day 15 up to Day 546 (Cohort 1) and Day 365 (Cohorts 2 and 3)
Geometric Mean Titer (GMT) of Histo-blood Group Antigen (HBGA)-blocking Antibodies Titers Against Vaccine Matched Genotypes | Day 1 and Day 29
Geometric Mean Fold Rise (GMFR) of HBGA-blocking Antibodies Titers Against Vaccine Matched Genotypes | Day 1 and Day 29
Percentage of Participants with Seroresponse Based on HBGA-blocking Antibody Titer | Day 29
GMT of Binding Antibody (bAb) Against Vaccine-matched NoV Genotypes | Day 1 and Day 29
GMFR of bAb Titers | Day 1 and Day 29
Percentage of Participants with Seroresponse Based on bAb Titer | Day 29

CONTACTS AND LOCATIONS:
Locations (281):
- United States (182):
  - Accel Research Sites - Achieve Clinical Research, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Alliance for Multispecialty Research, LLC, Daphne, Alabama
  - ClinMed, LLC, Phoenix, Arizona
  - DM Clinical - Phoenix, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Abby's Research Institute, Phoenix, Arizona
  - Headlands Research Scottsdale, Scottsdale, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Hope Research Institute - Tempe, Tempe, Arizona
  - Arizona Liver Health, Tucson, Arizona
  - Quality of Life Medical and Research Center, Tucson, Arizona
  - Del Sol Research Management LLC.- Tucson, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - ARK Clinical Research, LLC, Fountain Valley, California
  - ASCADA Research, LLC - Family Medicine, Fullerton, California
  - Matrix Clinical Research, Huntington Park, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Ark Clinical Research, Long Beach, California
  - Matrix Clinical Research, Los Angeles, California
  - Velocity Clinical Research - Westlake, Los Angeles, California
  - Paradigm Research, Redding, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Benchmark Research, Riverside, California
  - Peninsula Research Associates (PRA), Rolling Hills Estates, California
  - Apex Clinical Research, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Tekton Research - Fort Collins, Fort Collins, Colorado
  - Tekton Research, Inc - Longmont Center, Longmont, Colorado
  - Imagine Research of Palm Beach County, Boynton Beach, Florida
  - Pioneer Clinical Studies, Coral Gables, Florida
  - Integrity Clinical Research, LLC (ICR SITES) - Doral, Doral, Florida
  - Alliance for multispecialty Research - Florida, Doral, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Best Quality Research Inc., Hialeah, Florida
  - Neoclinical Research, Hialeah, Florida
  - Research Centers of America, Hollywood, Florida
  - Nature Coast Clinical Research, LLC - Inverness, Inverness, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Health Awareness INC, Jupiter, Florida
  - University Clinical Research- Deland, Lake Mary, Florida
  - Meridien Research, Lakeland, Florida
  - Clinical Site Partners - Leesburg, Leesburg, Florida
  - Accel Clinical Research - Maitland, Maitland, Florida
  - Dade Research Center, LLC, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Universal Axon Clinical Research, Miami, Florida
  - Florida International Research Center, Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Felicidad Medical Research, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - SUNCOAST Clinical Research, New Port Richey, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - United Medical Research, Port Orange, Florida
  - Health Awareness, Inc, Port Saint Lucie, Florida
  - St. Johns Center for Clinical Research, Saint Augustine, Florida
  - IMA Clinical Research - St. Petersburg, St. Petersburg, Florida
  - Global Clinical Professionals, LLC, St. Petersburg, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Albany Internal Medicine, Albany, Georgia
  - Delricht Research At Springer Wellness And Restorative Health, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CenExel iResearch Atlanta, LLC, Decatur, Georgia
  - Javara Inc., Fayetteville, Georgia
  - Fellows Research Alliance, Inc., Savannah, Georgia
  - Velocity Clinical Research-Savannah, Savannah, Georgia
  - Clinical Research Atlanta/Headlands, Stockbridge, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - IMA Clinical Research, Chicago, Illinois
  - Great Lakes Clinical Trials - Gurnee, Gurnee, Illinois
  - Bioluminix Clinical Research Chicago, Naperville, Illinois
  - Optimal Research, Peoria, Illinois
  - DM Clinical Research- River Forest, River Forest, Illinois
  - Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - Velocity Clinical Research-Sioux City, Sioux City, Iowa
  - Johnson County Clin-Trials (JCCT), Lenexa, Kansas
  - Velocity Clinical Research- Kansas City, Overland Park, Kansas
  - Tekton Research, Wichita, Kansas
  - AMR Lexington, Lexington, Kentucky
  - Velocity Clinical Research - Baton Rouge, Baton Rouge, Louisiana
  - Velocity Clinical Research - Covington, Covington, Louisiana
  - Benchmark Research, Metairie, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Privia Medical Group, Annapolis, Maryland
  - Cenexel CBH (CBH Health), Gaithersburg, Maryland
  - Velocity Clinical Research-Rockville, Rockville, Maryland
  - Javara Inc/Privia Medical Group, LLC, Silver Spring, Maryland
  - DM Clinical Research - Brookline, Brookline, Massachusetts
  - Skylight Health Research - Burlington, Burlington, Massachusetts
  - Headlands Research - Detroit, Southfield, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - DM Clinical Research - Southfield, Southfield, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Velocity Clinical Research, Gulfport, Gulfport, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Clinvest Headlands LLC, Springfield, Missouri
  - Delricht Research, Springfield, Missouri
  - Montana Medical Research, Inc, Missoula, Montana
  - Velocity Clinical Research-Lincoln, Lincoln, Nebraska
  - Velocity Clinical Research-Norfolk, Norfolk, Nebraska
  - Velocity Clinical Research-Omaha, Omaha, Nebraska
  - Javara Inc. / Nevada Health Centers, Ind, Carson City, Nevada
  - Vector Clinical Trials, Las Vegas, Nevada
  - Oasis Clinical Research, Las Vegas, Nevada
  - DM Clinical Research - New Jersey, Jersey City, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Albuquerque Clinical Trials (ACT), Albuquerque, New Mexico
  - DM Clinical Research, Albuquerque, New Mexico
  - Velocity Clinical Research- Albuquerque, Albuquerque, New Mexico
  - Velocity Clinical Research - Binghamton, Binghamton, New York
  - DM Clinical - Brooklyn, Brooklyn, New York
  - Brooklyn Clinical Research, Brooklyn, New York
  - Velocity Clinical Research - Syracuse, East Syracuse, New York
  - Drug Trials America, Hartsdale, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Velocity Clinical Research-Vestal, Vestal, New York
  - DelRicht Research, LLC, Charlotte, North Carolina
  - Javara Inc. - Tryon Medical-South Park, Charlotte, North Carolina
  - Velocity Clinical Research, Durham, Durham, North Carolina
  - West Clinical Research, Morehead City, North Carolina
  - Accellacare Raleigh, Raleigh, North Carolina
  - Accellacare of Wilmington, Wilmington, North Carolina
  - Javara - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Velocity Clinical Research, Cleveland, Beachwood, Ohio
  - Velocity Clinical Research-Mt. Auburn, Cincinnati, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Reseach - Blue Ash, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati OH, Cincinnati, Ohio
  - Centricity Research, Columbus, Ohio
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Tekton Research, Inc - Edmond, Edmond, Oklahoma
  - Delricht Tate, Tulsa, Oklahoma
  - Tekton Research, Inc - Yukon Location, Yukon, Oklahoma
  - Altoona Center for Clinical Research - Research, Duncansville, Pennsylvania
  - DM Clinical Research, Philadelphia, Pennsylvania
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Velocity Clinical Research - Anderson, Anderson, South Carolina
  - DelRicht Research, Charleston, South Carolina
  - Coastal Carolina Research Center - North Charleston, North Charleston, South Carolina
  - Velocity Clinical Research, Spartanburg, Spartanburg, South Carolina
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Delricht Moyer, Hendersonville, Tennessee
  - CNS Healthcare DBA Clinical Neuroscience Solutions, INC, Memphis, Tennessee
  - Benchmark Research, Austin, Texas
  - IMA Clinical Research Austin, Austin, Texas
  - Tekton Research, Inc. - Beaumont, Beaumont, Texas
  - Headlands Research Brownsville, Brownsville, Texas
  - Family Medicine Associates of Texas, Carrollton, Texas
  - Javara Inc (Conroe), Conroe, Texas
  - WR-Global Medical Research, LLC, Dallas, Texas
  - El Paso Research, El Paso, Texas
  - Benchmark Research, Fort Worth, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - DM Clinical Research - CyFair, Houston, Texas
  - DM Clinical Research - Bellaire, Houston, Texas
  - DM Clinical Research - Irving, Irving, Texas
  - ACRC Trials, Plano, Texas
  - Research Your Health, Plano, Texas
  - Delricht Research At Zomnir Family Medicine, Prosper, Texas
  - DM Clinical Research - San Antonio, San Antonio, Texas
  - IMA Clinical Research, San Antonio, Texas
  - Tekton Research Inc - San Antonio, San Antonio, Texas
  - DM Clinical Research - Sugarland, Sugar Land, Texas
  - DM Clinical Research - Tomball, Tomball, Texas
  - DM Clinical Research, Tomball, Texas
  - Cope Family Medicine, Bountiful, Utah
  - JBR Clinical Research, Salt Lake City, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Velocity Clinical Research - Hampton, Hampton, Virginia
  - Health Research of Hampton Roads, Newport News, Virginia
  - AMR Norfolk, Norfolk, Virginia
  - Velocity Clinical Research-Portsmouth, Portsmouth, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - DM Clinical Research - Seattle, Seattle, Washington
  - Frontier Clinical Research, LLC, Kingwood, West Virginia
- Australia (11):
  - Paratus Clinical Research Canberra, Bruce, Australian Capital Territory
  - Northside Health, Coffs Harbour, New South Wales
  - Momentum Clinical Research Darlinghurst, Darlinghurst, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Paratus Clinical Research Brisbane, Herston, Queensland
  - Griffith University Hospital, Southport, Queensland
  - Fusion Clinical Research, Norwood, South Australia
  - Veritus Research, Bayswater, Victoria
  - Emeritus Research (Melbourne), Camberwell, Victoria
  - The Peter Doherty Institute for Infection & Immunity, North Melbourne, Victoria
- Canada (19):
  - CARe Clinic, Calgary
  - Intermed Groupe Sante, Chicoutimi
  - Medicor Research Inc., Greater Sudbury
  - Apex Trials, Guelph
  - Isaak Walton Killam Health Centre, Halifax
  - Okanagan Clinical Trials, Kelowna
  - Centricity Research Quebec City, Lévis
  - Milestone Research Inc., London
  - Centricity Research Mirabel, Mirabel
  - Centricity Research Pointe-Claire, Pointe-Claire
  - Centre de Recherche Saint-Louis, Québec
  - Clinique Spécialisée en Allergie de la Capitale, Québec
  - CARe Clinic Red Deer, Red Deer
  - Richmond Clinical Trials, Richmond
  - Bluewater Clinical Research Group, Inc, Sarnia
  - Diex Research Sherbrooke Inc, Sherbrooke
  - Centricity Research Toronto LMC, Toronto
  - Diex Recherche Trois-Rivières, Trois-Rivières
  - Colchester Research Group, Truro
- Japan (23):
  - Chubu Rosai Hospital - Rheumatology & Collageous, Nagoya, Aichi-ken
  - Daido clinic, Nagoya, Aichi-ken
  - Medical Corporation JR Hiroshima Hospital, Hiroshima, Hirosima [Hiroshima]
  - Kotoni Medical Support Clinic, Sapporo, Hokkaidô [Hokkaido]
  - Tenjin Sogo Clinic, Fukuoka, Hukuoka [Fukuoka]
  - Matsuba Clinic, Kawasaki-shi, Kanagawa
  - Hayashi-Katagihara Clinic, Kyoto, Kyôto [Kyoto]
  - Yokoi Medicine Clinic, Minoh, Osaka
  - Asano Clinic, Kawagoe-shi, Saitama
  - Omi Medical Center, Yabasecho, Shiga
  - Dojinkinenkai Meiwa Hospital, Chiyoda-ku, Tôkyô [Tokyo]
  - Nihonbashi Sakura Clinic, Chūōku, Tôkyô [Tokyo]
  - Medical Corporation Asbo Tokyo Asbo Clinic, Minatoku, Tôkyô [Tokyo]
  - Tokyo Saiseikai Central Hospital, Minatoku, Tôkyô [Tokyo]
  - Denenchofu Family Clinic, Ōta-ku, Tôkyô [Tokyo]
  - Higashi-Shinjuku Clinic - Internal Medicine, Shinjuku-ku, Tôkyô [Tokyo]
  - Shimamura Memorial Hospital, Suginami City, Tôkyô [Tokyo]
  - P-one Clinic, Hachiōji, Tôkyô
  - Sasaki Clinic, Hyōgo
  - NewHeart Watanabe Institute, Kanazawa
  - Izumino Hospital, Kochi
  - Sapporo Odori Endoscopy Clinic, Sapporo
  - Takatsuki General Hosiptal, Takatsuki-shi
- Panama (4):
  - CEVAXIN David, David, Chiriquí Province
  - CEVAXIN Chorrera, La Chorrera
  - CEVAXIN 24 de Diciembre, Panama City
  - CEVAXIN Avenida Mexico, Panama City
- Puerto Rico (3):
  - BRCR Global, Ponce
  - Clinical Research Puerto Rico, Inc., San Juan
  - Research Works San Juan, San Juan
- United Kingdom (39):
  - Velocity Clinical Research - High Wycombe, High Wycombe, Buckinghamshire
  - Warrington and Halton Teaching Hospitals NHS Foundation Trust - Halton General Hospital, Runcorn, Cheshire
  - Royal Cornwall Hospitals NHS Trust - Royal Cornwall Hospital, Truro, Cornwall
  - St George's University Hospitals NHS Foundation Trust - St George's Hospital, London, England
  - Accellacare South London, Orpington, Kent
  - Layton Medical Centre, Blackpool, Lancashire
  - Panthera Biopartners - Manchester, Rochdale, Manchester
  - Northern Care Alliance NHS Foundation Trust - Salford Royal Hospital, Salford, Manchester
  - Lakeside Healthcare, Corby, Northamptonshire
  - Eynsham Medical Center, Witney, Oxfordshire
  - NHS Grampian - Aberdeen Royal Infirmary, Aberdeen
  - NIHR Welcome Trust Clinical Research Facility, Birmingham
  - Bournemouth Research Hub, Bournemouth
  - North Bristol NHS Trust - Southmead Hospital, Bristol
  - Cardiff and Vale University Health Board - University Hospital Wales, Cardiff
  - Accellacare Warwickshire Quality Research Site, Coventry
  - NHS Lothian - Western General Hospital, Edinburgh
  - Panthera Biopartners - North London, Enfield
  - Royal Devon & Exeter Hospital (Wonford), Exeter
  - CPS Research by FutureMeds, Glasgow
  - Glasgow Clinical Research Facility, Glasgow
  - Panthera Biopartners - Glasgow, Glasgow
  - University Hospitals of Leicester NHS Trust, Leicester
  - FutureMeds Wirral, Liverpool
  - Mile End Hospital, London
  - Royal Free London NHS Foundation Trust - Royal Free Hospital, London
  - Manchester University NHS Foundation Trust, Manchester
  - FutureMeds Newcastle, Newcastle upon Tyne
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Leeds Teaching Hospitals NHS Trust - St James' University Hospital, Nottingham
  - Plymouth Hospital NHS trust-Derriford Hospital, Plymouth
  - Portsmouth Research Hub, Portsmouth
  - Panthera Biopartners - Sheffield, Sheffield
  - Accellacare Yorkshire Quality Research Site, Shipley
  - Wansford Research Ltd, Wansford
  - Weymouth Research Hub, Weymouth
  - Windrush Medical Practice, Witney
  - North Wales Clinical Research Centre (NWCRC), Wrexham
  - Panthera Biopartners - York, York